CLINICAL TRIAL: NCT04636840
Title: Leveraging Social Media to Identify and Connect Teens With Eating Disorders to a Mobile Guided Self-Help Mobile Intervention
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); SilverCloud Health (Unknown); Palo Alto University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH119170-01 (NIH)
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Eating Disorders
Keywords: mHealth; eating disorders; bulimia nervosa; binge eating disorder; teens; adolescents; social media
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Control Group (No Intervention): Access to a self-help version of Space From Body and Eating Concerns Program on SilverCloud Health App
- Experimental Group A- Mobile App with Social Networking Feature (Experimental): Access to a coached Space From Body and Eating Concerns program on SilverCloud Health App with private social media group for social networking support.
  Interventions: Device: Space From Body and Eating Concerns- Teen
- Experimental Group B- Mobile App Only (Experimental): Access to a coached Space From Body and Eating Concerns program on SilverCloud Health App.
  Interventions: Device: Space From Body and Eating Concerns- Teen

INTERVENTIONS:
Device: Space From Body and Eating Concerns- Teen — Mobile application with coaching component
  Arms: Experimental Group A- Mobile App with Social Networking Feature; Experimental Group B- Mobile App Only

SUMMARY:
Clinical or subclinical eating disorders (EDs) impact 10% of individuals in their lifetime and are marked by significant functional impairment, early mortality, chronicity, and emotional distress. ED symptoms often emerge in adolescence, with peak onset age in the teenage years. Early recognition and treatment of these devastating illnesses are needed to prevent long-term consequences and a chronic course. Most (80%) individuals with EDs, including teens with EDs (TwEDs), do not receive treatment. Due to major barriers to access and to the delivery of treatment for TwEDs, there is a need for a new model of service delivery that can identify and help TwEDs. We demonstrated our ability to harness social media to identify and efficiently recruit large numbers of TwEDs. Our team has successfully developed a guided self-help cognitive behavioral therapy (CBT)-based mobile app for previous studies and have adapted this app to address the specific needs of TwEDs. In proposed study, we will test this updated mHealth intervention, which includes simplified language and tailored content relevant to adolescent issues and a social networking feature designed to facilitate group exchanges. This mHealth intervention will be investigated among 161 TwEDs recruited from Instagram/Facebook to test preliminary efficacy and feasibility of this mHealth intervention to improved eating disorder symptoms among TwEDs not currently engaged in treatment. We will also garnering feedback via a mixed methods approach on the efficiency, technical effectiveness, and satisfaction with mHealth intervention content and features. Participants will be randomized to one of 3 study arms, including a control group (self-help version of the app), a group with access to the coached mobile app only, and a group with access to the coached mobile app plus social networking feature. We hypothesized that those with access to the coached mobile app intervention will have improved ED outcomes in comparison to the control group, and that those with access to the additional social networking feature will have the most improvement in ED symptoms out of all three groups.

ELIGIBILITY:
Inclusion Criteria:

* US Resident
* Owns or has daily access to an iOS or Android smartphone
* English-speaking
* Screen Positive for a DSM-5 subclinical/clinical eating disorder other than anorexia nervosa (AN) or at high risk for an eating disorder

Exclusion Criteria:

* Currently Engaged in eating disorder treatment
* Screen Positive for Anorexia Nervosa
* Wards of the State or Foster Children

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 161 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Symptoms | Baseline, 6 weeks, 3 months, 6 months
  Change of eating disorder symptoms as evaluated by the Eating Disorders Examination Questionnaire (EDE-Q) global score.

SECONDARY OUTCOMES:
Quality of Life Scores | Baseline, 6 weeks, 3 months, 6 months
  Change in quality of life scores among participants will be evaluated using the Pediatric Quality of Life Short Form (PedsQL 4.0).
Utilization/Uptake of Treatment | Baseline, 6 weeks, 3 months, and 6 months
  Uptake of mental health treatment will include beginning treatment in participants' assigned condition (i.e., uptake of version of app to which they were assigned) or receipt of any other treatment type (i.e., in-person).

OTHER OUTCOMES:
Depression Symptoms | Baseline, 6 weeks, 3 months, 6 months
  Change in depression symptoms as evaluated by the Pediatric Health Questionnaire for Adolescents (PHQ-A).
Anxiety Symptoms | Baseline, 6 weeks, 3 months, 6 months
  Change in depression symptoms as evaluated by the Screen for Child Anxiety Related Disorders (SCARED).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be deidentified and uploaded into data sharing structures on the NIMH Data Archive as compliant with funding source requirements.
Time Frame: Summary data will be available on NIMH Data Archive as compliant with funding source requirements.
Access Criteria: Summary data will be available on NIMH Data Archive as compliant with funding source requirements.